CLINICAL TRIAL: NCT04576559
Title: Effect of Modified Dental Visual Aids on Behavior Management During Dental Treatment in Children With Autism Spectrum Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Abdulaziz University (Other)
Responsible Party: Principal Investigator, Ala Aljubour, Principal Investigator, King Abdulaziz University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: KingAbdulazizUni
Record Dates: First submitted 2020-09-30; First posted 2020-10-06 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Child Autism
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified dental visual aids (Experimental)
  Interventions: Other: Modified dental visual aids
- Regular dental visual aids (Active Comparator)
  Interventions: Other: Regular dental visual aids

INTERVENTIONS:
Other: Modified dental visual aids — Modified Dental visual aids in the form of pictures created by the main investigator
  Arms: Modified dental visual aids
Other: Regular dental visual aids — Regular dental visual aids
  Arms: Regular dental visual aids

SUMMARY:
There is a need to find an approach that is appropriate for managing children with Autism Spectrum Disorder in the dental clinic, to manage their behaviour and decrease their anxiety in this research we will apply our modified dental visual aids and test its effectiveness in managing the behavior of such children during the dental appointment.

ELIGIBILITY:
Inclusion Criteria:

* Patient age between 6-10 years.
* Child patient has to represent the typical triad symptoms of ASD that include: social interaction deficits, communication impairment, language impairment and rigidity of interests.
* Child patient with ASD diagnosis confirmed in the patient's files according to "the DSM-V criteria" (American Psychiatric Association, 2013).
* Child patient with mild to moderate ASD according to "the Childhood Autism Rating Scale (CARS)" (Schopler et al., 1998).

Exclusion Criteria:

* Patient age younger than 6 years and older than 10 years.
* Child patient with other congenital anomalies, for example, "Cerebral Palsy" or "Down Syndrome".
* Child patient with previous dental experience.
* Child patient with severe ASD according to "the Childhood Autism Rating Scale (CARS)" (Schopler et al., 1998).

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Plaque Index Scoring | four weeks
  plaque index scoring (Silness and Löe, 1964)
Anxiety Scale for Children with Autism Spectrum Disorder (ASC-ASD) | four weeks
  This scale contains twenty-four "self-report" questions that inquire about anxiety, it contains 4 sub-scales including:
  1. Separation Anxiety (SA).
  2. Uncertainty (U).
  3. Performance Anxiety (PA).
  4. Anxious Arousal (AA). It is a four-point "Likert-scale"; items in the questionnaire are rated from zero ("never") to three ("always"). Another version of the same scale with twenty-four questions directed to the parents will also be used and it contains a report of their child's symptoms of anxiety, within the same four subscales (Rodgers et al., 2016).
The Observational Scale of Behavioral Distress (OSBD) | four weeks
  This scale is used to measure the behavioral distress that a child experiences when undergoing a painful procedure. This scale is composed of eight operationally defined behaviors that are indicative of anxiety and/or pain behavior in children. The OSBD is a valid and reliable scale that measures distress in children receiving painful procedures in the medical and dental practice, for example, venipuncture and needle injections (Elliot et al., 1987).

CONTACTS AND LOCATIONS:
Locations (1):
- King Abdulaziz University, Jeddah, Select A State Or Province, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No